CLINICAL TRIAL: NCT03549000
Title: A Phase I/Ib, Open-label, Multi-center, Study of NZV930 as a Single Agent and in Combination With PDR001 and/or NIR178 in Patients With Advanced Malignancies.
Brief Title: A Phase I/Ib Study of NZV930 Alone and in Combination With PDR001 and /or NIR178 in Patients With Advanced Malignancies.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After review of data which showed low likelihood of efficacy in these patients Novartis decided to terminate the trial early. Termination was not safety related
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNZV930X2101; 2018-000153-51 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Triple Negative Breast Cancer (TNBC); Pancreatic Ductal Adenocarcinoma (PDAC); Colorectal Cancer Microsatellite Stable (MSS); Ovarian Cancer; Renal Cell Carcinoma (RCC); Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: NZV930; PDR001; NIR178; Immune checkpoint inhibitor; immunotherapy; CD73; PD-1; PD-L1; A2aR; Adenosine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell | interventions — Biological Products; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NZV930 Monotherapy (Experimental): Single Agent NZV930
  Interventions: Other: NZV930
- NZV930 with PDR001 Doublet Therapy (Experimental): Combination of NZV930 with PDR001
  Interventions: Other: NZV930; Other: PDR001
- NZV930 with NIR178 Doublet Therapy (Experimental): Combination of NZV930 with NIR178
  Interventions: Other: NZV930; Drug: NIR178
- NZV930 with NIR178 & PDR001 Triplet Therapy (Experimental): Combination of NZV930 with NIR178 and PDR001
  Interventions: Other: NZV930; Other: PDR001; Drug: NIR178

INTERVENTIONS:
Other: NZV930 — NZV930, Specified dose on specified days, intravenous (IV)
  Other Names: Biological
Other: PDR001 — PDR001, Specified dose on specified days, intravenous (IV)
  Other Names: Biological
  Arms: NZV930 with NIR178 & PDR001 Triplet Therapy; NZV930 with PDR001 Doublet Therapy
Drug: NIR178 — NIR178 Specified dose on specified days, Orally
  Arms: NZV930 with NIR178 & PDR001 Triplet Therapy; NZV930 with NIR178 Doublet Therapy

SUMMARY:
The purpose of this study was to assess the safety, tolerability, and preliminary anti-tumor activity of experimental medication NZV930 alone and when combined with PDR001 and/or NIR178, in patients with advanced cancers

ELIGIBILITY:
Inclusion Criteria:

Adult men & women ≥ 18 years of age Histologically confirmed advanced malignancies with documented progression following standard therapy, or for whom, in the opinion of the investigator, no appropriate standard therapy exists.

Must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. The patient must be willing to undergo a new tumor biopsy at screening and during treatment.

ECOG performance status 0-2 and in the opinion of the investigator, likely to complete at least 56 days of treatment.

Exclusion Criteria:

Symptomatic or uncontrolled Brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.

Patients with treated symptomatic brain metastases should be neurologically stable for 4 weeks post-treatment prior to study entry and at doses of <10 mg per day prednisolone or equivalent for at least 2 weeks before administration of any study treatment.

Patients who required discontinuation of treatment due to treatment-related toxicities with prior immunotherapy.

Patients previously treated with anti-CD73 treatment and/or adenosine receptor A2a (A2aR) inhibitors.

Active, previously documented, or suspected autoimmune disease within the past 2 years.

Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur should not be excluded. Additionally, patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.

History of or current drug-induced interstitial lung disease or pneumonitis grade ≥ 2.

Impaired cardiovascular function or clinically significant cardiovascular disease, including any of the following: Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2), uncontrolled hypertension or clinically significant arrhythmia Patients with corrected QT using the Fridericia's correction (QTcF) > 470 msec for females or >450 msec for males, on screening ECG or congenital long QT syndrome Acute myocardial infarction or unstable angina < 3 months prior to study entry History of stroke or transient ischemic event requiring medical therapy Symptomatic claudication Infection: HIV infection, Active HBV or HCV infection (per institutional guidelines). Patients with chronic HBV or HCV disease that is controlled under antiviral therapy are allowed in the expansion but not in the escalation, Known history of tuberculosis Infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed treatment before screening is initiated.

Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 6 weeks is indicated as washout period. For patients receiving anticancer immunotherapies, 4 weeks is indicated as the washout period.

Systemic chronic steroid therapy (≥ 10 mg/day prednisone or equivalent) or any immunosuppressive therapy, other than replacement dose steroids in the setting of adrenal insufficiency, within 7 days of the first dose of study treatment. Topical, inhaled, nasal, and ophthalmic steroids are allowed

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of the NZV930 in combination with PDR001 and/or NIR178 | 3 years
  Incidence and severity of AEs and SAEs, incl. changes in laboratory parameters, vital signs, and ECGs Dose limiting toxicity in cycle 1 (28 days) for single agent NZV930 and NZV930 in combination with PDR001 and/or NIR178 during dose escalation phase only Tolerability: dose interruptions Tolerability: dose reductions Tolerability: dose intensity

SECONDARY OUTCOMES:
Overall response rate (ORR) | 3 years
  Defined as the proportion of patients with best overall response of CR or PR
Clinical Benefit Rate (CBR) | 3 years
  Defined as the proportion of patients with best overall response of CR, PR or SD >= 16 weeks
Progression Free Survival (PFS) | 3 years
  Defined as the time from the date of start of treatment to the date of the event defined as first documented progression or death due to any cause
Serum concentration vs. time profiles of NZV930 (free drug) and PDR001. | 3 years
  Serum concentration vs. time profiles of NZV930 (free drug) and PDR001.
Plasma concentration vs. time profiles for NIR178 and derived PK parameters | 3 years
  Concentration time profile of NIR178 and its metabolites
To assess the immunogenicity of NZV930 and PDR001 | 3 years
  Presence and titer of anti-drug antibodies, anti-NZV930 and anti-PDR001 in (patients receiving combination with PDR001).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (2):
  - H Lee Moffitt Cancer Center and Research Institute Inc, Tampa, Florida
  - University of Texas MD Anderson Cancer Center MD Anderson PSC, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18104
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1879